CLINICAL TRIAL: NCT04955535
Title: Screening of Specific Genes for Pigmented Villous Nodular Synovitis
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M201947901
Record Dates: First submitted 2021-06-25; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Pigmented Villonodular Synovitis
MeSH Terms: conditions — Synovitis, Pigmented Villonodular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Arthroscopic synovectomy — Arthroscopic synovectomy

SUMMARY:
This study retrospectively analyzed the history of present illness of PVNS patients in our hospital. The enrolled patients were followed up by telephone to follow up their postoperative recovery and living conditions. Take the patient's pathological specimens for immunohistochemical testing, evaluate the relationship between the expression of different molecular targets, clinical manifestations and patient prognosis, and explore new molecular targets related to disease diagnosis and treatment.

DETAILED DESCRIPTION:
This study retrospectively analyzed the symptoms, time of onset, injury history, laboratory examinations, imaging examinations, and intraoperative conditions of PVNS patients in our hospital. The enrolled patients were followed up by telephone to follow up their postoperative recovery and living conditions (VAS score, SF-36 score). Take the patient's pathological specimens for immunohistochemical testing, evaluate the relationship between the expression of different molecular targets, clinical manifestations and patient prognosis, and explore new molecular targets related to disease diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of pigmented villonodular synovitis.
2. Clinical diagnosis of giant cell tumor of tendon sheath

Exclusion Criteria:

1. No surgical treatment.
2. There were no pathological specimens during the operation.
3. The age of the patient is less than 18 years old or more than 60 years old.
4. The operation record shows nodular type.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with "pigmented villonodular synovitis" and "giant cell tumor of tendon sheath"
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2020-12-27 (Actual); Study Completion 2020-12-27 (Actual)

PRIMARY OUTCOMES:
Difference of scale score between immunohistochemistry positive group and negative group | One week after surgery
  Difference of Visual Analog Score for pain between CSF-1 immunohistochemistry positive group and negative group
Difference of Visual Analog Score for pain between TNF-α immunohistochemistry positive group and negative group | One week after surgery
  Difference of Visual Analog Score for pain between TNF-α immunohistochemistry positive group and negative group
Difference of Visual Analog Score for pain between IL-1B immunohistochemistry positive group and negative group | One week after surgery
  Difference of Visual Analog Score for pain between IL-1B immunohistochemistry positive group and negative group
Difference of SF-36 score between CSF-1 immunohistochemistry positive group and negative group | One week after surgery
  Difference of SF-36 score between CSF-1 immunohistochemistry positive group and negative group
Difference of SF-36 score between TNF-α immunohistochemistry positive group and negative group | One week after surgery
  Difference of SF-36 score between TNF-α immunohistochemistry positive group and negative group
Difference of SF-36 score between IL-1B immunohistochemistry positive group and negative group | One week after surgery
  Difference of SF-36 score between IL-1B immunohistochemistry positive group and negative group

SECONDARY OUTCOMES:
Correlation between basic demographic characteristics and scale scores | One week after surgery
  Correlation between age, gender and scale score

CONTACTS AND LOCATIONS:
Overall Officials: Yingfang Ao, Prof., Study Chair — Peking Yniversity Third Hospital
Locations (1):
- Institute of Sports Medicine, Peking University Third Hospital, Beijing Key Laboratory of Sports Injuries， Beijing, China, Beijing, Beijing Municipality, China